CLINICAL TRIAL: NCT04723771
Title: Influenza Vaccination Effectiveness of a Quadrivalent Inactivated Vaccine in Pregnant Women and Young Infants (Aged 6 Months and Below) During Influenza Season 2019/2020
Brief Title: Influenza Vaccine Effectiveness of a Quadrivalent Vaccine in Pregnant Women and Young Infants, 2019-2020
Status: Completed | Type: Observational
Sponsor: University of Athens (Other)
Collaborators: Hellenic Pasteur Institute (Unknown)
Responsible Party: Principal Investigator, Helena Maltezou, Professor, University of Athens
Other Study IDs: 16708
Record Dates: First submitted 2020-09-22; First posted 2021-01-26 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Influenza in Human
Keywords: influenza; quadrivalent influenza vaccine; influenza vaccine effectiveness; pregnancy; pregnant women; infants
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Influenza is associated with an increased risk for serious illness, hospitalization and death in pregnant women and young infants. The investigators estimated the effectiveness of a quadrivalent inactivated influenza vaccine (QIV) in pregnant women and their infants in 2019-2020 influenza season. Women were activelly followed during the influenza season on a weekly basis through telephone call in order to collect data about the onset of fever and/or respiratory symptoms by them or their young infants. Polymerase chain reaction testing in pharyngeal samples was offered to pregnant women and infants with influenza-like illness (ILI). A total of 636 pregnant women and 474 infants were studied. A Bayesian beta-binomial model was used.

DETAILED DESCRIPTION:
Study period: Influenza 2019-2020 season

The investigators followed actively the pregnant women and their infants in order to collect prospectively data on a weekly basis through phone calls during the entire influenza season.

Definitions:

* ILI was defined as the sudden onset of symptoms and fever, malaise, myalgia or headache, and cough, sore throat or shortness of breath.
* ARI was defined as the presence of at least one respiratory symptom, regardless of fever.
* Febrile episode was defined as the presence of fever only.
* Fever was defined as a temperature of 38.0 C in at least two measurements within 24h.
* The diagnoses of pneumonia and AOM were accepted as reported by the physicians who provided care to the women or their infants.

The 2019-2020 QIV Vaxigrip-Tetra was used to vaccinate pregnant women.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women >18 years old and <45 years old, cared at Alexandra General Hospital (Athens, Greece) between October 16 and January 27, 2020

Exclusion Criteria:

* <18 years old or >45 years old
* not in stable health
* already vaccinated against influenza
* history of Guillain-Barré syndrome
* history of hypersensitivity to influenza vaccines
* immunosuppression
* history of investigational drug <30 days
* history of immunoglobulins or blood products <3 months
* fever at day of interview (enrollment day)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women and their infants
Sampling Method: Non-Probability Sample
Enrollment: 949 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
rates of laboratory-confirmed influenza in vaccinated and unvaccinated pregnant women | 2019-2020 influenza season
  influenza vaccine effectiveness against laboratory-confirmed influenza in pregnant women
rates of laboratory-confirmed influenza in young infants whose mothers were vaccinated and in infants of unvaccinated mothers | 2019-2020 influenza season
  influenza vaccine effectiveness against laboratory-corfirmed influenza in young infants

SECONDARY OUTCOMES:
rates of acute respiratory infection, influenza-like illness, febrile episode, use of antibiotics, use of antivirals, pneumonia, acute otitis media (for infants only), healthcare seeking and hospitalization in pregnant women and their infants | 2019-2020 influenza season
  influenza vaccine effectiveness against the abovementioned secondary outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Loutradis, Professor, Principal Investigator — First Department of Obstetrics and Gynecology, University of Athens
Locations (1):
- First Department of Obstetrics and Gynecology, University of Athens, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided
In order to share IPD we should request permission from the Ethics Committee of the hospital.

REFERENCES:
- [Derived] Maltezou HC, Stavros S, Asimakopoulos G, Pergialiotis V, Raftopoulos V, Talias MA, Pavli A, Daskalakis G, Sindos M, Koutroumanis P, Theodora M, Antsaklis P, Kostis E, Stratiki E, Kossyvakis A, Theodoridou M, Mentis A, Drakakis P, Loutradis D, Rodolakis A. Effectiveness of maternal vaccination with quadrivalent inactivated influenza vaccine in pregnant women and their infants in 2019-2020. Expert Rev Vaccines. 2022 Jul;21(7):983-992. doi: 10.1080/14760584.2022.2013820. Epub 2022 Jan 24. PMID 34878959

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/71/NCT04723771/SAP_001.pdf